CLINICAL TRIAL: NCT06973421
Title: Preliminary Phase II Clinical Study on the Efficacy and Safety of the Combination of Utidelone Capsules and Fruquintinib Capsules in the Treatment of Platinum Resistant Recurrent Ovarian Cancer
Brief Title: Phase II Study of Utidelone Plus Fruquintinib Combination Therapy for Platinum-Resistant Recurrent Ovarian Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xiaohua Wu MD [zzhong], Professor, Director of Gynecologic Oncology, Fudan University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FRUTD-001
Record Dates: First submitted 2025-05-07; First posted 2025-05-15 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Platinum Resistant Ovarian Cancer
MeSH Terms: interventions — HMPL-013

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Utidelone+Fruquintinib (Experimental): Participants will receive Utidelone Capsules and Fruquintinib Capsules in combination. 21 days as a cycle.
  Interventions: Drug: Utidelone Capsules; Drug: Fruquintinib Capsules

INTERVENTIONS:
Drug: Utidelone Capsules — 60 mg/m2 orally, days 1 to 5, per cycle
Drug: Fruquintinib Capsules — 5 mg orally, days 1 to 14, per cycle

SUMMARY:
This study is a Prospective, Single-arm, Phase 2 clinical trial. The purpose of this study is to find out if taking Utidelone Capsules together with Fruquintinib Capsules is safe and works well for people with platinum-resistant ovarian cancer . Researchers will look at the Objective Response Rate, Progression-Free Survival, Overall Survival, safety, and any side effects.

ELIGIBILITY:
Inclusion Criteria:

1. The subjects were fully informed, voluntarily signed the informed consent, and were willing and able to follow the planned visit, research treatment plan, laboratory examination and other research procedures.
2. Female subjects aged ≥ 18 and ≤ 70 at the time of signing the informed consent.
3. Malignant epithelial ovarian cancer, fallopian tube cancer or primary peritoneal cancer were confirmed by histology or pathology.
4. Subjects had at least one measurable lesion defined by RECIST v1.1.
5. The number of lines of previous systematic anti-tumor treatment ≤ 3 (neoadjuvant and adjuvant chemotherapy are not considered as previous systematic treatment, unless disease progression occurs during its chemotherapy or within 6 months after the last chemotherapy).
6. ECoG physical status score was 0 or 1.
7. The baseline examination confirmed that there was sufficient bone marrow and organ function, and no relevant supportive treatment, such as gcs-f, EPO or blood transfusion, was used within 14 days before the laboratory examination in the screening period. (see the table on the next page for specific indicators)
8. The expected survival time was more than 12 weeks.
9. Fertile patients must agree to use reliable contraceptive methods (hormone or barrier method or abstinence) with their partners during the trial and at least 3 months after the last medication; The blood or urine pregnancy test of female patients of childbearing age must be negative before enrollment.

Exclusion Criteria:

1. It has clear cell, mucinous or sarcomatous histology, contains mixed tumors of any histological type, or low-grade/borderline ovarian cancer.
2. In platinum refractory ovarian cancer subjects, platinum refractory was defined as the best response during the first platinum containing regimen treatment as disease progression or recurrence, or disease recurrence or progress within 4 weeks after the end of platinum containing regimen treatment.
3. Other malignant tumors within 5 years, excluding cured basal cell carcinoma of the skin, carcinoma in situ of the cervix and papillary carcinoma of the thyroid.
4. Received nitrosourea or mitomycin C within 6 weeks before the first use of the study drug; received anti-tumor treatment within 4 weeks or 5 half lives (whichever is shorter) before the first use of the study drug, including chemotherapy, radiotherapy, biological targeted therapy, immunotherapy, etc; Oral fluorouracil, small molecule targeted drugs and endocrine therapy were used 2 weeks before the first use of the study drug or within 5 half lives of the drug (whichever is shorter); Traditional Chinese medicine or Chinese patent medicine with anti-tumor indications were used within 2 weeks before the first use of the study drug.
5. Major surgical operations (craniotomy, thoracotomy or laparotomy or other operations defined by the investigator) or significant trauma were performed within 60 days before the first use of the study drug, or elective surgery was required during the trial.
6. There were patients with clinically significant skin wounds, surgical sites, wound sites, severe mucosal ulcers or fractures that were not completely healed as assessed by the researchers.
7. Patients with peripheral neuropathy with CTCAE 5.0 rating ≥ 2.
8. The adverse reactions of previous anti-tumor treatment have not recovered to CTCAE 5.0 grade evaluation ≤ 1 (except for the toxicity without safety risk judged by researchers such as hair loss).
9. Patients who have previously received eutidylon or antiangiogenic drugs (except bevacizumab).
10. Urine protein detection 2+or more, or 24-hour urine protein quantitation ≥ 1.0g/24h.
11. There were symptoms or thyroid dysfunction requiring treatment at the time of screening.
12. Patients with obvious evidence of bleeding tendency or medical history within 2 months before the first use of the study drug, such as black stool, hematemesis, hemoptysis, occult blood in stool++, etc.
13. Subjects with active central nervous system metastasis.
14. Cancerous ascites with clinical symptoms requiring puncture and drainage; Or those who received drainage for the purpose of treatment within 30 days before the first use of the study drug.
15. During screening, it was found that the tumor invaded the structure of large blood vessels, such as pulmonary artery, superior vena cava or inferior vena cava, and the researchers judged that there was a high risk of bleeding; Or there is a history of previously known aneurysms.
16. There was a history of arterial thrombosis or deep venous thrombosis within 6 months before the first use of the study drug; Thrombosis caused by implantable venous infusion pump or catheter, or superficial venous thrombosis, except those with stable thrombosis after regular anticoagulation therapy.
17. Patients with coagulation disorders, bleeding tendency, or undergoing anticoagulation therapy 2 months before the first use of the study drug.
18. Have a history of serious cardiovascular and cerebrovascular diseases, including but not limited to:

    Acute myocardial infarction, severe/unstable angina pectoris or coronary artery bypass grafting within 6 months before the first use of the study drug; The New York Heart Association (NYHA) classification of congestive heart failure was ≥ 2; LVEF<50%； Or there is a history of myocarditis (including patients who have been cured after treatment of previous myocarditis) or other grade 3 or above cardiovascular events; Stroke events and/or transient cerebral ischemia occurred within 12 months before the first use of the study drug; Patients with uncontrolled hypertension (systolic blood pressure ≥ 140 mmHg or diastolic blood pressure ≥ 90 mmHg) were given standard treatment; Other researchers judged that there was a high risk of heart disease.
19. Uncontrolled diabetic patients within 3 months before the first use of the study drug.
20. Patients with active hepatitis B and/or C, i.e. HBsAg positive and/or HBcAb positive, detected HBV DNA positive and/or anti HCV positive and HCV RNA positive at the same time; Human immunodeficiency virus (HIV) antibody was positive; Treponema pallidum specific antibody was positive.
21. active infection or fever of unknown origin (body temperature>38.5 ℃) before screening and first use of the study drug.
22. patients with active autoimmune diseases need systemic treatment (i.e. disease regulators, corticosteroids or immunosuppressive drugs) within 2 years before enrollment. Replacement therapy (such as thyroxine, insulin or physiological corticosteroid replacement therapy for adrenal or pituitary insufficiency) is not considered as a systemic treatment.
23. women who are pregnant or nursing or plan to be pregnant during the study period.
24. patients with mental disorders or poor compliance.
25. known allergic to the study drug or any of its excipients.
26. participate in another intervention clinical trial or use other research treatment at the same time.
27. the researcher believes that the subject has a serious history of systemic diseases or other reasons and is not suitable to participate in the trial.

Ages: 18 Years to 75 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-07-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
ORR | Up to 24 months
  Objective response rate, according to RECIST v1.1

SECONDARY OUTCOMES:
CA-125 remission rate | Up to 24 months
  evaluated according to gcic CA-125 standard
PFS | approximately 2 years
  Progression-free survival, according to RECIST v1.1
OS | Up to 2 years
  Overall survival, according to RECIST v1.1
AEs | From the first drug administration to within 30 days for the last treatment dose
  Adverse Events, according to CTCAE V5.0 criteria, During the trial, the adverse event record form should be truthfully filled in, including the occurrence time, severity, correlation with study treatment, duration, measures taken and outcome of the adverse event.

CONTACTS AND LOCATIONS:
Locations (1):
- Fudan University Shanghai Cancer Cente, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided
Data is available per require after approved by ethics broad